CLINICAL TRIAL: NCT05915338
Title: The Eof ıInsulin Use Education on Safe Drug Administration, Pain Level and Perception of Treatment in Patients With Type 2 Diabetes
Brief Title: Training on Using ıInsulin in Patients With Type 2 Diabetes
Acronym: İNSÜLİN
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Serap Parlar Kılıç, Professor Doctor, Inonu University
Other Study IDs: INONU UNİV
Record Dates: First submitted 2023-06-09; First posted 2023-06-23 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Insulin Dependent Diabetes; Diabetes type2
Keywords: Tip 2 Diyabet; Güvenli İlaç Kullanımı; Tedavi Algısı; İnsülin
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: -Pre-test data were obtained by using the descriptive information form, İUBGF, VAS, and HRAS.
  The patients were asked to self-administer a dose of insulin that day, and the ability of the patients to administer the insulin dose was recorded in the IUBGF as the 1st follow-up by the researchers. Afterwards, individual insulin use training was given and the "Educational Manual on the Use of Insulin for Individuals with Type 2 Diabetes" was given to the patients and the first follow-up was completed.
  -2 weeks later, post-test data were obtained from the patients using IUBGF, VAS, and HRAS. The ability of the patients to administer the insulin dose was recorded in the IUBGF as the second follow-up by the researchers.
  After 8 weeks, post-test data were obtained by using IUBGF, VAS, and HRAS as retention tests. The ability of the patients to administer the insulin dose was recorded by the researchers as the 3rd follow-up retention test in IUBGF.
- Control Group: -Pre-test data were obtained by using the descriptive information form, İUBGF, VAS, and HRAS.
  The patients were asked to self-administer a dose of insulin that day, and the ability of the patients to administer the insulin dose was recorded in the IUBGF as the 1st follow-up by the researchers.
  -2 weeks later, post-test data were obtained from the patients using IUBGF, VAS, and HRAS. Patients were asked to self-administer a daily dose of insulin. The ability of the patients to administer the insulin dose was recorded in the IUBGF as the second follow-up by the researchers.
  After 8 weeks, post-test data were obtained by using IUBGF, VAS, and HRAS as retention tests. Patients were asked to self-administer a daily dose of insulin. The ability of the patients to administer the insulin dose was recorded in IUBGF as the 3rd follow-up retention test by the researchers.

SUMMARY:
This study was conducted to evaluate the effect of individual insulin use training given to patients with type 2 diabetes using insulin on safe drug administration, pain level and perception of treatment. The study was conducted between October 2022 and March 2023 with a randomized control group.

DETAILED DESCRIPTION:
Objective: The aim of this study was to examine the effects of individual insulin use training given to patients with Type 2 diabetes on safe drug administration, pain level and treatment perception, and to contribute to both national and international literature.

Method: It was conducted between October 2022 and March 2023 as a randomized controlled study in a pre-test-post-test order to determine the effect of individual insulin use education given to patients with type 2 diabetes on safe drug administration, pain level and treatment perception. The data were collected by the researchers with the descriptive information form of the patients, the Insulin Administration Skill Observation Form, the Visual Analogue Scale and the Insulin Therapy Evaluation Scale.

Data Collection: Face-to-face and individual interviews with patients who applied to the Internal Diseases and Endocrinology Polyclinic and Diabetes Nursing Polyclinics of a state hospital in a city located in the Southeastern Anatolia Region of Turkey, and who were hospitalized in the Internal Diseases, Endocrinology, Physical Therapy and Rehabilitation and Cardiology Services. collected using the method. A pilot study was not conducted before starting the study. Before the study, all patients were informed about the study and their verbal and written consents were obtained.

ELIGIBILITY:
Inclusion Criteria:

Patients included in the study;

* 18 years and over Using insulin injections for at least six months or longer
* Meeting the American Diabetes Association (ADA, 2021) diagnostic criteria for Type 2 diabetes
* No communication and mental problems
* Insulin injection made by himself or his family The patients who agreed to participate in the study.

Exclusion Criteria:

Patients excluded from the study;

* Self or family member health personnel Those with advanced retinopathy, nephropathy, neuropathy
* Diagnosed with type 1 diabetes
* Pregnant or breastfeeding women
* Patients who participated in another clinical trial concurrently or within 1 month prior to the start of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 Diabetes
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Fırst follow - up survey | Fırst test-fırst applıcatıon both groups at the begınnıng of the research
  Pretest data was obtained using the introductory information form, IASOF, VAS, and ITES.
  Patients were requested to apply their daily dose of insulin to themselves and patients' application skills were recorded by the researchers into IASOF as the 1st observation.

SECONDARY OUTCOMES:
Last test survey | 2 weeks after the fırst watch
  Posttest data was obtained through the use of IASOF, VAS, and ITES. Patients were requested to apply their insulin dose of the day to themselves. Patients' insulin application skills were recorded by researchers into IASOF as the 2nd observation.

OTHER OUTCOMES:
Durabılıty test for both groups | After 8 weeks, the follow-up test was done to both groups
  Posttest data was obtained through the use of IASOF, VAS, and ITES. Patients were requested to apply their insulin dose of the day to themselves. Patients' insulin application skills were recorded by researchers into IASOF as the 3rd observation.

CONTACTS AND LOCATIONS:
Locations (1):
- Şirnak Devlet Hastanesi, Şirnak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozturk MH, Kerkez M, Kilic SP. The power of insulin education: enhancing pain and treatment perception in adult type 2 diabetes patients. J Diabetes Metab Disord. 2025 Jun 5;24(1):140. doi: 10.1007/s40200-025-01652-2. eCollection 2025 Jun. PMID 40485759